CLINICAL TRIAL: NCT00571441
Title: Estimating Volume Using LiDCO Versus Other Measures of Volume
Brief Title: Estimating Volume Using LiDCO
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00002786
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2009-03

CONDITIONS: Brain Injury; Ischemic Stroke; Hemorrhagic Stroke
Keywords: stroke; Brain injury; nursing; Critical care
MeSH Terms: conditions — Brain Injuries; Ischemic Stroke; Hemorrhagic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: All subjects are included in this group, non-randomized observational study.

SUMMARY:
We hypothesize that the stroke volume variation measured using the commercially available LiDCO monitor provides a reasonable estimate of volume when compared to standard measures. This study will collate data that is already being collected by the bedside nurses.

DETAILED DESCRIPTION:
Objective: To compare measurement of stroke volume variance with intake/output measurements, weight, BUN/Creatnine values, and central venous pressure.

Design: Non-experimental, non-randomized observational comparative study.

Setting: The sixteen bed Neurocritical Care Unit at Duke University Hospital.

Patients: 45 adult (over 18 years) subjects with intracranial pathology who require volume resuscitation. Only patients with current LiDCO monitoring will be considered eligible for inclusion in the study.

Interventions: This is an observational study. Subjects will receive standard-of-care treatment without additional intervention.

Data Analysis: All data will be collected by the principal investigator / study coordinator. Personal patient information will be removed (deidentified) from the permanent data collection records to protect patient confidentiality. Data collected will be entered into a Microsoft Excel electronic spreadsheet and will be saved on a USB Disk drive to be stored in a locked cabinet in the investigator's office. Statistical analysis using SAS v9.1, (Cary, NC) will be conducted with a level of significance set at .05 (alpha) using standardized comparative analysis techniques.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the neurocritical care unit have an arterial line in place already connected to LiDCO monitor Physician order for monitoring intake and output

Exclusion Criteria:

* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurologically injured patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Stroke volume variation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai Olson, PhD RN CCRN, Study Director — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Pearse RM, Ikram K, Barry J. Equipment review: an appraisal of the LiDCO plus method of measuring cardiac output. Crit Care. 2004 Jun;8(3):190-5. doi: 10.1186/cc2852. Epub 2004 May 5. PMID 15153237
- [Background] Linton RA, Jonas MM, Tibby SM, Murdoch IA, O'Brien TK, Linton NW, Band DM. Cardiac output measured by lithium dilution and transpulmonary thermodilution in patients in a paediatric intensive care unit. Intensive Care Med. 2000 Oct;26(10):1507-11. doi: 10.1007/s001340051347. PMID 11126264